CLINICAL TRIAL: NCT04361396
Title: Assessment of the Presence of the SARS-COV-2 Virus in the Peritoneum During an Emergency Laparoscopy Conducted on Confirmed or Suspected COVID-19 Patients
Brief Title: Assessment of the Presence of the SARS-COV-2 Virus in the Peritoneum of COVID-19 Patients
Acronym: LAPTRANSCOV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHRD 0420
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2022-05

CONDITIONS: Coronavirus Infection
Keywords: Emergency laparoscopy; Coronavirus Infections; SARS-CoV-2; pneumoperitoneum; COVID-19
MeSH Terms: conditions — Coronavirus Infections; Pneumoperitoneum; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Collection of samples (Other): Only in enrolled patient : different samples will be taken at different times of the surgery (3 samples of pneumoperitoneum, 1 sample of peritoneal effusion or peritoneal lavage fluid and 1 sample of bile, in case of cholecystectomy).
  Interventions: Other: Collection of samples

INTERVENTIONS:
Other: Collection of samples — Only in enrolled patient : different samples will be taken at different times of the surgery (3 samples of pneumoperitoneum, 1 sample of peritoneal effusion or peritoneal lavage fluid and 1 sample of bile, in case of cholecystectomy.

SUMMARY:
The purpose of this study is to determine whether the virus SARS-CoV-2, responsible for the disease COVID-19, is present in the abdominal cavity during emergency laparoscopic exploration in confirmed or suspected COVID-19 patients.

DETAILED DESCRIPTION:
A new human coronavirus responsible for pneumonia, SARS-CoV-2, emerged in China in December 2019 and has spread rapidly worlwide. COVID-19, the disease caused by this virus, has a very polymorphous clinical presentation, which ranges from upper respiratory tract infections to acute respiratory distress syndrome. Research institutions are working restlessly to elucidate the physiopathology of COVID-19 to develop new and more efficacious strategies on diagnosis, treatment and prevention planning. However, many aspects of the disease process are still unknown. Despite the lack of complete understanding of COVID-19, recommandations from world health authorities to surgical societies have been published in order to prevent viral transmission within the hospital setting. Concerning prevention of viral transmission during laparoscopy on confirmed or suspected COVID-19 cases, strict measures were taken to protect surgical and anesthesia staff. These recommandations are mainly based on avoiding leak of pneumoperitoneum during surgical exploration as it may represent a potential source of viral transmission, eventhough there is no scientific evidence on it. The lack of evidence of this mode of transmission makes difficult to develop more appropriate and efficacious recommandations. This study is designed to assess for the presence of SARS-CoV-2 virus in the peritoneal serosa during emergency laparoscopy on confirmed or suspected COVID-19 cases. During laparoscopic surgical exploration, 3 samples of pneumoperitoneum will be taken in 3 standardized steps of the procedure. Two more other samples of peritoneal effusion or peritoneal lavage (in the absence of peritoneal effusion) and bile (if cholecystectomy is performed) will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Patient COVID-19 diagnosed by positive RT-PCR SARS-CoV-2 for less than 10 days, or by thorax CT-scan suggesting specificdiagnostic aspects of COVID-19 requiring abdominal or gynecological surgery by emergency laparoscopy

OR

* Patient COVID-19 suspected requiring abdominal or gynecological surgery by emergency laparoscopy. Suspicion will be defined by the presence of at least one of the following symptoms:
* Cough for less than 15 days
* Fever which appeared recently and which excluded another etiology
* Anosmia without obstructive rhinitis
* Contact with a COVID-19 + case person less than 21 days ago
* Patient requiring abdominal or gynecological surgery by emergency laparoscopy and who should be tested by RT-PCR SARS-CoV-2
* Written and signed consent of the patient or guardian or family or, if this is not possible, emergency inclusion procedure
* Patients with affiliation to French social security system

Exclusion Criteria:

* Patient already participating in research involving the human person
* Negative RT-PCR SARS-CoV-2
* Withdrawal of patient or guardian or family; or refusal to sign the required inform consent form to continue to participate in the Clinical Trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
Assessment of the presence of the SARS-COV-2 virus at T4 | After surgery, an average of half a day
  Assessment of the presence of the SARS-COV-2 virus by RT-PCR in the peritoneum at the end of the surgical procedure with exsufflation (T4) in COVID-19 patients

SECONDARY OUTCOMES:
Assessment of the presence of the SARS-COV-2 virus at T1 | After surgery, an average of half a day
  Assessment of the presence of the SARS-COV-2 virus by RT-PCR immediately after creation of the pneumoperitoneum just before intraperitoneal surgical exploration (T1) in COVID-19 patients
Assessment of the presence of the SARS-COV-2 virus in the peritoneal effusion at T2 or T4 | After surgery, an average of half a day
  Assessment of the presence of the SARS-COV-2 virus by RT-PCR in the peritoneal effusion found during surgical exploration (T2) or in the peritoneal lavage fluid at the end of the surgical procedure before exsufflation (T4) in COVID-19 patients
Assessment of the presence of the SARS-COV-2 virus at T3 | After surgery, an average of half a day
  Assessment of the presence of the SARS-COV-2 virus by RT-PCR in the pneumoperitoneum during intraperitoneal surgical dissection (T2) with straight blunt/sharp or any kind of energy devices in COVID-19 patients
Assessment of the presence of the SARS-COV-2 virus at T5 | After surgery, an average of half a day
  Assessment of the presence of the SARS-COV-2 virus by RT-PCR in the bile at the end of the intervention after specimen extraction (T5), in case a cholecystectomy is performed in COVID-19 patients

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Trelles, Principal Investigator — Hôpital NOVO
Locations (5):
- France (5):
  - CH Victor Dupouy, Argenteuil
  - CH Intercommunal, Créteil
  - Department of General and Digestive Surgery, Hospital René Dubos, Pontoise
  - Department of Gynecology-Obstetrics, Hospital René Dubos, Pontoise
  - CH Delafontaine, Saint-Denis